CLINICAL TRIAL: NCT04840251
Title: Investigating the Feasibility of a Randomised Controlled Trial of a Physiotherapy Well-being Review in Patients With Pulmonary Hypertension.
Brief Title: Investigating a Well-being Review in Pulmonary Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH20898
Record Dates: First submitted 2021-03-23; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Pulmnary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): The treatment group will have a physiotherapy well-being review and be referred for rehabilitation. They will be seen after 6 months for follow-up
  Interventions: Other: Well-being review and rehabiliation
- Control (No Intervention): The control group will have initial assessments then receive brief advice on exercise. They will also be followed up after 6 months
- Qualitative (Other): to understand how it feels to take part in the well-being review, we will interview some participants who have already had this kind of treatment and ask questions about their experiences of it and how it was for them. We are also interested to know what differences they felt it made so that we can help to decide about the things we want to measure as outcomes in the interventional of the study.
  Interventions: Other: Qualitative Interviews

INTERVENTIONS:
Other: Well-being review and rehabiliation — For their well-being review, patients will meet with a physiotherapist specialist in PH and discuss:
  * how they are
  * what they can do for themselves
  * what it is challenging for them to do
  * how active they are
  * if they have ever exercised before The physiotherapist will then make a referral to the most suitable rehabilitation service local to the patient e.g. rehabilitation classes, physiotherapy at home, weight-loss programmes.
  Arms: Intervention
Other: Qualitative Interviews — Patients who have previously undergone rehabilitation will take part in a semi-structured interview to explore their experience and the impact it has had
  Arms: Qualitative

SUMMARY:
Pulmonary Hypertension (PH) is a rare disease that makes patients easily become breathless. There is evidence that people with PH can benefit from exercise; we want to look at how they can access rehabilitation in their local community.

Aim: To see if it is feasible to study physiotherapy well-being reviews in PH. Step 1: We will interview some patients with PH who have had rehabilitation and ask questions about their experiences. We will also ask what they think we should measure to show any difference their rehabilitation has made to them. The findings from Step 1 will help us to shape the details of Step 2, where we will conduct a small study to see if it is feasible to run a full study. Participants will be divided randomly into a treatment group and a control group. The treatment group will have a physiotherapy well-being review, leading to referral to their most suitable local rehabilitation service and follow-up after 6 months. The control group will receive brief exercise advice and follow-up after 6 months. The findings will help to design a full study and be shared with patients and health professionals.

ELIGIBILITY:
Inclusion Criteria:

* in World Health Organisation (WHO) Functional Class II or III
* have a diagnosis of PH
* have started on PH drug therapy in the preceding 18 months
* showing no signs of worsening breathlessness or heart failure
* on an unchanged PH therapeutic regime for at least 6 months prior to inclusion.

Exclusion Criteria:

* have an active infection or acute exacerbation of lung disease
* have participated in a clinical study involving another investigation of drug, device or exercise within the previous 6 months
* are on a surgical or other pathway of care that has pre-determined physiotherapy or activity regimes or restrictions
* have any additional medical conditions that may adversely affect the safety of the subject or severely limit the lifespan of the subject
* have participated in rehabilitation in the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
6MWD | Follow up at 6 months
  Change from Baseline in how far he patient can walk in 6 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Sospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No